CLINICAL TRIAL: NCT01143766
Title: Premedication With Single Dose Gabapentin to Improve Patient Tolerance in ERCP: A Double-Blind Randomized Controlled Trial
Brief Title: Gabapentin to Improve Patient Tolerance in Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Gregory A. Cote, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0911-51
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Conscious Sedation
Keywords: Sedation; Gabapentin; ERCP; Endoscopy
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard sedation (Active Comparator): Patients will receive combination opiate and benzodiazepine for sedation, the current standard of care.
  Interventions: Other: Standard sedation regimen
- Gapabentin (Active Comparator): Patients will receive gabapentin 900mg PO x 1 dose, one hour prior to the procedure. At the time of ERCP, patients will be sedated in a standard fashion.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — gabapentin 900mg PO x 1 dose, 1 hour prior to the procedure
  Arms: Gapabentin
Other: Standard sedation regimen — Combination opiate and benzodiazepine will be administered to achieve moderate sedation. This is the standard of care.
  Arms: Standard sedation

SUMMARY:
The standard approach to sedation in endoscopic retrograde cholangiopancreatography (ERCP) involves the use of benzodiazepines and opiates to achieve a moderate depth of sedation. There is data to suggest supplementing this regimen with gabapentin may lead to reduced pain, higher patient satisfaction and lower opiate requirements. The investigators are conducting a clinical trial to study this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age referred to IUMC for first-time ERCP procedure.

Exclusion Criteria:

1. Pregnant women
2. age <18 years
3. Incarcerated individuals
4. Patients currently taking or having taken gabapentin or pregabalin within the last 3 months
5. Patients unable to give informed consent
6. Patients not able to fill out visual analog scales for pain, nausea and anxiety or unable to fill out survey regarding procedural satisfaction.
7. High risk patients for anesthesia: home oxygen, class III or IV heart failure, sleep apnea (on CPAP/BiPAP at home), or ASA class > 3.
8. Patients undergoing general anesthesia for their ERCP procedure
9. Patients receiving propofol sedation for their ERCP procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Cote, MD, MS, Principal Investigator — Indiana University
Locations (1):
- University Hospital, Indiana University Purdue University Indianapolis, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Sedation | Gapabentin
Started | 25 | 31
Completed | 25 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Sedation | Gapabentin | Total
Number analyzed (Participants) | 25 | 31 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 27 | 48
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (16.6) | 48.1 (12.8) | 48.6 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 25 | 31 | 56

OUTCOME MEASURES:

1. Primary Outcome: Dosing Requirements
Description: Assess the effect of a single 900mg dose of gabapentin pre- ERCP on intra and post procedure narcotic/sedative requirements.
Time Frame: At time of discharge post-procedure
Population: TOTAL DOSE OF MEPERIDINE
Measure: Median (Inter-Quartile Range); unit: TOTAL DOSE OF MEPERIDINE, mg
Arm/Group | Standard Sedation | Gapabentin
Number analyzed (Participants) | 25 | 31
TOTAL DOSE OF MEPERIDINE, mg | 100 [88 to 125] | 100 [100 to 150]

2. Secondary Outcome: Number of Participants With Sedation-Related Adverse Events
Description: Sedation-related adverse events
Time Frame: At time of discharge post-procedure
Measure: Number; unit: participants
Arm/Group | Standard Sedation | Gapabentin
Number analyzed (Participants) | 25 | 31
participants | 3 | 2

3. Secondary Outcome: Median Pain Score at Time of Discharge
Description: Assess the effect of a single 900mg dose of gabapentin on pain at time of discharge, measured by a visual analog scale ranging from 0 (worst pain) to 100 (no pain).
Time Frame: At time of discharge post-procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Sedation | Gapabentin
Number analyzed (Participants) | 25 | 31
units on a scale | 80 [39 to 100] | 95 [87 to 100]

4. Secondary Outcome: Median Anxiety Score at Time of Discharge
Description: Assess the effect of a single 900mg dose of gabapentin on anxiety at time of discharge, measured by a visual analog scale ranging from 0 (worst anxiety) to 100 (no anxiety).
Time Frame: At time of discharge post-procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Sedation | Gapabentin
Number analyzed (Participants) | 25 | 31
units on a scale | 99 [95 to 100] | 98 [94 to 100]

5. Secondary Outcome: Median Nausea Score at Time of Discharge
Description: Assess the effect of a single 900mg dose of gabapentin on nausea at time of discharge, measured by a visual analog scale ranging from 0 (worst nausea) to 100 (no nausea).
Time Frame: At time of discharge post-procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Sedation | Gapabentin
Number analyzed (Participants) | 25 | 31
units on a scale | 99 [92 to 100] | 95 [84 to 100]

ADVERSE EVENTS:
Arm/Group | Standard Sedation | Gapabentin
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/31
Other Adverse Events (participants affected / at risk) | 3/25 | 4/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Sedation (N=25) | Gapabentin (N=31)
Hypoxemia or apnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 0 | 2 (2)

LIMITATIONS AND CAVEATS:
Limited sample size due to challenges with recruitment and transition to propofol-based anesthesia for sedation in ERCP. Study terminated at 50% enrollment for this reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No